CLINICAL TRIAL: NCT02214407
Title: A Randomized Phase III Study of Decitabine (DAC) With or Without Hydroxyurea (HY) Versus HY in Patients With Advanced Proliferative Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Randomized Phase III Study of Decitabine +/- Hydroxyurea (HY) Versus HY in Advanced Proliferative CMML
Acronym: GFM-DAC-CMML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-DAC-CMML
Record Dates: First submitted 2014-07-30; First posted 2014-08-12 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: MDS
MeSH Terms: interventions — Decitabine; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A: DECITABINE (DACOGEN) (Experimental): Decitabine (DAC) will be administered at 20 mg/m2 intravenously daily for 5 days every 28 days.
  Allopurinol, 300mg/d, will be started at the time of inclusion; hydration during treatment will be administered to all patients. In (the rare) case of necessity, prophylactic anti-emetics could be given.
  Hydroxyurea may be added during the first 3 cycles if WBC counts > 30 G/L, and mandatory if WBC > 50 G/L. The daily dose will be adapted to maintain WBC below 15 to 20 G/L.
  Interventions: Drug: Decitabine
- ARM B: HYDROXYUREA (Experimental): Hydroxyurea (HY) 1g/d once daily, with dose adjustments (up to 4g/d) to maintain a WBC count between 5 and 10 G/L. Allopurinol, 300mg/d started at the time of inclusion will be administered to all patients.
  Dose escalation will be performed by steps of 0.5 g/d, up to 4 g/d, if the WBC has been reduced by less than 20% and remains > 15 G/L. HY will then be adapted to maintain a WBC count between 5 and 10 G/L. HY will be lowered if platelets decrease by > 30 X 109/L (if initially below 100 X 109L). HY will be discontinued in cases of grade 4 thrombocytopenia or neutropenia, and reintroduced at a lower dose after recovery to grade ≤ 3. Persistent grade 4 thrombocytopenia or neutropenia after a 4 week discontinuation will mandate bone marrow evaluation.
  Interventions: Drug: HYDROXYUREA

INTERVENTIONS:
Drug: Decitabine — Decitabine (DAC) will be administered at 20 mg/m2 intravenously daily for 5 days every 28 days. Hydroxyurea may be added during the first 3 cycles if WBC counts > 30 G/L, and mandatory if WBC > 50 G/L. The daily dose will be adapted to maintain WBC below 15 to 20 G/L.
  Treatment will be continued until an event is reached. Events and thus study exit will be acknowledged only after agreement between the investigator and a Trial Committee.
  Other Names: DACOGEN
  Arms: ARM A: DECITABINE (DACOGEN)
Drug: HYDROXYUREA — Hydroxyurea (HY) 1g/d once daily, with dose adjustments (up to 4g/d) to maintain a WBC count between 5 and 10 G/L. Allopurinol, 300mg/d started at the time of inclusion will be administered to all patients.
  Treatment will be continued until an event is reached. Events and thus study exit will be acknowledged only after agreement between the investigator and a Trial Committee.
  Arms: ARM B: HYDROXYUREA

SUMMARY:
This is a phase III, two-arm, randomized, stratified, multicenter, open-label study with individual therapeutic benefit aim:

Decitabine (DAC) with or without Hydroxyurea (HY) versus HY in patients with advanced proliferative Chronic Myelomonocytic Leukemia (CMML)

The primary objective of the study is to compare between the two arms Event-free Survival (EFS).

Secondary objectives are to compare between both arms:

Overall Survival (OS) Cumulative incidence of AML Overall and Complete Response Rates at 3 and 6 cycles according to IWG 2006 criteria modified for CMML Response duration Toxicity (hematological and non hematological) Prognostic factors

DETAILED DESCRIPTION:
ARM A: DECITABINE (DAC)

Decitabine (DAC) will be administered at 20 mg/m2 intravenously daily for 5 days every 28 days.

Treatment will be delayed at the discretion of the investigator (up to D56) for febrile neutropenia (≥ 38.5°C; absolute neutrophil count [ANC], < 1,000/μL), clinical and/or microbiologic infection with grade 3 to 4 neutropenia (ANC < 1,000/μL), or hemorrhage with grade 4 thrombocytopenia (< 25,000 platelets/μL). If renal or hepatic dysfunction occurs, treatment will be stopped until resolution or withheld if dysfunction persists more than 4 days. Persistent grade 4 thrombocytopenia or neutropenia beyond D49 will mandate bone marrow evaluation.

Treatment will be continued until an event is reached. Events and thus study exit will be acknowledged only after agreement between the investigator and a Trial Committee.

Allopurinol, 300mg/d, will be started at the time of inclusion; hydration during treatment will be administered to all patients. In (the rare) case of necessity, prophylactic anti-emetics could be given.

Hydroxyurea may be added during the first 3 cycles if WBC counts > 30 G/L, and mandatory if WBC > 50 G/L. The daily dose will be adapted to maintain WBC below 15 to 20 G/L.

ARM B: HYDROXYUREA (HY)

Hydroxyurea (HY) 1g/d once daily, with dose adjustments (up to 4g/d) to maintain a WBC count between 5 and 10 G/L. Allopurinol, 300mg/d started at the time of inclusion will be administered to all patients.

Treatment will be continued until an event is reached. Events and thus study exit will be acknowledged only after agreement between the investigator and a Trial Committee. This is intended to prevent early dropout, notably in the HY arm.

Dose escalation will be performed by steps of 0.5 g/d, up to 4 g/d, if the WBC has been reduced by less than 20% and remains > 15 G/L. HY will then be adapted to maintain a WBC count between 5 and 10 G/L. HY will be lowered if platelets decrease by > 30 X 109/L (if initially below 100 X 109L). HY will be discontinued in cases of grade 4 thrombocytopenia or neutropenia, and reintroduced at a lower dose after recovery to grade ≤ 3. Persistent grade 4 thrombocytopenia or neutropenia after a 4 week discontinuation will mandate bone marrow evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* CMML diagnosis according to WHO criteria Stable excess in blood monocytes, > 1 G/L Lack of bcr-abl rearrangement (or Philadelphia chromosome) Bone marrow blast cells < 20% Dysplasia of at least one lineage or clonality marker or blood monocytosis during more than 3 months w/o other explanation Blood and marrow smears will be reviewed at each country's level, but morphologist meetings at the 3 country level are planned for better harmonization and review of difficult cases
* WBC ≥ 13 G/L Measured on two successive CBC at least two weeks apart, outside of a context of infection.
* Either D1 or D2

D1: At least two of the following criteria, reviewed at each country's level: (modified from Wattel et al. Blood 1996) Marrow blasts >= 5 % Clonal cytogenetic abnormality (other than t(5;12) (q33; p13) and isolated loss of Y chromosome ) Anemia (Hb < 10 g/dL) ANC > 16 G/l (in absence of infection) Thrombocytopenia (platelet count < 100 G/L) Splenomegaly > 5 cm below costal margin (spleen size should also be measured by an imaging technique)

Or:

D2: Extramedullary involvement: Including documented cutaneous, pleural or pericardial effusion.

* No prior treatment (except supportive care, or ESA, or short term (< 6 weeks) HY in patients presenting with high WBC counts)
* Performance status 0-2 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Adequate organ function including the following Hepatic : total bilirubin < 1.5 times upper limit of normal (ULN) (except moderate unconjugated hyperbilirubinemia due to intra medullary hemolysis or Gilbert syndrome) , alanine transaminase (ALT) and aspartate transaminase (AST) < 3xULN Renal : serum creatinine < 2 x ULN
* Signed Informed consent
* Negative pregnancy and adequate contraception (including in male patients wishing to father) if relevant.

Exclusion Criteria:

* Myeloproliferative / myelodysplastic syndrome other than CMML
* CMML with t(5 ;12) or PDGFBR rearrangement that may receive imatinib
* Patients eligible for allogeneic bone marrow transplantation with an identified donor
* Pregnant or breastfeeding
* Performance status > 2 on the ECOG Scale.
* Serious concomitant systemic disorder, including active bacterial, fungal or viral infection that in the opinion of the investigator would compromise the safety of the patient and/or his/her ability to complete the study
* Prior malignancy (except in situ cervix carcinoma, limited basal cell carcinoma, or other tumors if not active during the last 3 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
compare between the two arms Event-free Survival (EFS) | 3 months
  Comparison of Event-free Survival between both arms. Events will include
  * Death from any cause
  * Disease Progression, defined as one of the following: (i) at any time point: transformation to AML according to WHO criteria ; (ii) after at least 6 cycles of treatment: doubling of bone marrow blasts to > 10%, and worsening of cytopenias lasting for > 4 weeks ; (iii) after at least 3 cycles of treatment: Progression of myeloproliferation (despite maximal HY or DAC dosing; in the absence of concomitant infection) defined as: ≥ 50% increase in spleen size as determined by an imaging technique or doubling in WBC or occurrence of a previously undiagnosed extramedullary localization of the disease.

SECONDARY OUTCOMES:
Overall Survival (OS) | 7 month
  Overall survival compared between both Arm of treatment (decitabine and hydroxyurea)
Cumulative incidence of AML | 7 month
  Comparaison of Cumulative incidence of AML between both arm of treatment (decitabine and hydroxyurea)
Overall and Complete Response Rates | 3 month
  Overall and Complete Response Rates at 3 and 6 cycles according to IWG 2006 criteria modified for CMML
Response duration | 3 month
  Comparison of response duration after 3 month and 6 month of treatment between both arm of treatment (decitabine and hydroxyurea)
Toxicity | 1 month
  hematological and non hematological
Prognostic factors | 3 month
  Prognostic factors of Event Free Survival with decitabine and hydroxyurea

CONTACTS AND LOCATIONS:
Overall Officials: ITZYKSON Raphael, PHD, Principal Investigator — Hopital Saint-Louis, Service hematologie Senior
Locations (45):
- France (45):
  - CHU La Réunion - Site nord, Saint-Denis, La Réunion
  - CHU La Réunion-Site Sud, Saint-Pierre, La Réunion
  - Chu Amiens, Amiens
  - CHU d'Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - Ch Avignon, Avignon
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hôpital Nord Franche-Comté, Belfort
  - Hôpital Avicenne, Bobigny
  - CHU de Brest - Hôpital Morvan, Brest
  - CHU Côte de Nacre, Caen
  - Hôpital privé Sévigné, Cesson-Sévigné
  - CHU Estaing, Clermont-Ferrand
  - CH de Compiègne, Compiègne
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Centre Henri Mondor, Créteil
  - CHU Albert Michallon, Grenoble
  - CH Le Mans, Le Mans
  - Clinique Victor Hugo, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - CHRU de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut Paoli-Calmette, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Clinique Beausoleil, Montpellier
  - Hôpital Saint Eloi, Montpellier
  - Hopital de l'Hotel Dieu, Nantes
  - Hopital Archet I, Nice
  - CHU de Nîmes, Nîmes
  - CHR d'Orléans, Orléans
  - Hopital St Louis T4, Paris
  - Centre Hospitalier Joffre, Perpignan
  - CHU de Haut-Lévèque, Pessac
  - CHU Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - CH Annecy Genevois, Pringy
  - CHU de Reims, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Bequerel, Rouen
  - Hôpital Hautepierre, Strasbourg
  - IUCT Oncopole - Département d'hématologie, Toulouse
  - Iuct Oncopole, Toulouse
  - CH Valence, Valence
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Institut gustave Roussy, Villejuif

REFERENCES:
- [Derived] Itzykson R, Santini V, Thepot S, Ades L, Chaffaut C, Giagounidis A, Morabito M, Droin N, Lubbert M, Sapena R, Nimubona S, Goasguen J, Wattel E, Zini G, Torregrosa Diaz JM, Germing U, Pelizzari AM, Park S, Jaekel N, Metzgeroth G, Onida F, Navarro R, Patriarca A, Stamatoullas A, Gotze K, Puttrich M, Mossuto S, Solary E, Gloaguen S, Chevret S, Chermat F, Platzbecker U, Fenaux P. Decitabine Versus Hydroxyurea for Advanced Proliferative Chronic Myelomonocytic Leukemia: Results of a Randomized Phase III Trial Within the EMSCO Network. J Clin Oncol. 2023 Apr 1;41(10):1888-1897. doi: 10.1200/JCO.22.00437. Epub 2022 Dec 1. PMID 36455187
- [Derived] Pleyer L, Leisch M, Kourakli A, Padron E, Maciejewski JP, Xicoy Cirici B, Kaivers J, Ungerstedt J, Heibl S, Patiou P, Hunter AM, Mora E, Geissler K, Dimou M, Jimenez Lorenzo MJ, Melchardt T, Egle A, Viniou AN, Patel BJ, Arnan M, Valent P, Roubakis C, Bernal Del Castillo T, Galanopoulos A, Calabuig Munoz M, Bonadies N, Medina de Almeida A, Cermak J, Jerez A, Montoro MJ, Cortes A, Avendano Pita A, Lopez Andrade B, Hellstroem-Lindberg E, Germing U, Sekeres MA, List AF, Symeonidis A, Sanz GF, Larcher-Senn J, Greil R. Outcomes of patients with chronic myelomonocytic leukaemia treated with non-curative therapies: a retrospective cohort study. Lancet Haematol. 2021 Feb;8(2):e135-e148. doi: 10.1016/S2352-3026(20)30374-4. PMID 33513373